CLINICAL TRIAL: NCT00001596
Title: Therapeutic Clinical Trial of Oral Pirfenidone for the Pulmonary Fibrosis of Hermansky-Pudlak Syndrome
Brief Title: Oral Pirfenidone for the Pulmonary Fibrosis of Hermansky-Pudlak Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: William Gahl, M.D. (NIH)
Collaborators: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor-Investigator, William Gahl, M.D., Clinical Director, National Human Genome Research Institute, National Human Genome Research Institute (NHGRI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 970085; 97-HG-0085
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Results first posted 2012-01-26 (Estimated); Last update posted 2017-10-16 (Actual); Status verified 2017-09

CONDITIONS: Albinism; Inborn Errors of Metabolism; Oculocutaneous Albinism; Platelet Storage Pool Deficiency; Pulmonary Fibrosis
Keywords: Albinism; Platelet Storage Pool Deficiency; Pulmonary Fibrosis; Hermansky-Pudlak Syndrome
MeSH Terms: conditions — Albinism; Metabolism, Inborn Errors; Albinism, Oculocutaneous; Platelet Storage Pool Deficiency; Pulmonary Fibrosis; Hermanski-Pudlak Syndrome | interventions — pirfenidone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pirfenidone (Active Comparator): Subjects received pirfenidone 801 mg (3 pills of 267 mg each), three times daily.
  Interventions: Drug: Pirfenidone
- Placebo (Placebo Comparator): Subjects received placebo (3 pills), three times daily.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pirfenidone — Treatment with pirfenidone 801 mg (3 pills of 267 mg each), three times daily.
  Other Names: Deskar; Esbriet
  Arms: Pirfenidone
Drug: Placebo — Placebo (3 pills), three times daily.
  Other Names: Inactive matching placebo
  Arms: Placebo

SUMMARY:
Hermansky-Pudlak Syndrome (HPS) is an inherited disease that results in decreased pigmentation (oculocutaneous albinism), bleeding problems due to a platelet abnormality (platelet storage pool defect), and storage of an abnormal fat-protein compound (lysosomal accumulation of ceroid lipofuscin).

The disease can cause poor functioning of the lungs, intestine, kidneys, or heart. The most serious complication of the disease is pulmonary fibrosis and typically causes death in patients 40 - 50 years old. The disorder is common in Puerto Rico, where many of the clinical research studies on the disease have been conducted. Neither the full extent of the disease nor the basic cause of the disease is known. There is no known treatment for HPS.

The drug pirfenidone blocks the biochemical process of inflammation and has been reported to slow or reverse pulmonary fibrosis in animal systems.

In this study researchers will select up to 40 HPS patients diagnosed with pulmonary fibrosis. The patients will be randomly divided into 2 groups. The patients will not know if they are taking pirfenidone or a placebo "sugar pill".

1. Group one will be patients who will receive pirfenidone.
2. Group two will be patients who will receive a placebo "sugar pill"

The major outcome measurement of the therapy will be a change in the lung function (forced vital capacity). The study will be stopped if one therapy proves to be more effective than the other.

DETAILED DESCRIPTION:
Hermansky-Pudlak Syndrome (HPS) is a rare autosomal recessive disease consisting of oculocutaneous albinism and a platelet storage pool defect. The most serious complication of this disorder, which is common in Puerto Rico, is pulmonary fibrosis, generally fatal in the fourth or fifth decade. There is no treatment for the pulmonary disease of HPS, which resembles idiopathic pulmonary fibrosis. However, a drug called pirfenidone has antifibrotic effects in animal models of lung fibrosis. Pirfenidone is an IND drug initially provided by Marnac, Inc.; InterMune, Inc., now holds the license. Pirfenidone inhibits cytokine-induced inflammation. Reported side effects include gastrointestinal upset, a photosensitivity rash, and palpitations. Between 1997 and 2001, we performed a randomized, placebo-controlled trial under this protocol that found pirfenidone to be safe and efficacious when analyzed using a repeated measures model. Using a random coefficients model, however, the data were definitive only in the restricted group of subjects whose initial forced vital capacity was greater than 50% of predicted. Because the repeated measures analysis had been chosen a priori as the optimal model, the DSMB stopped the study and directed that all patients receive pirfenidone. (Of the 23 original patients, 3 are still receiving pirfenidone under this protocol.)

Now, to prove efficacy of pirfenidone, we are conducting a block-randomized, placebo-controlled, double-blind trial involving up to 40 HPS patients whose forced vital capacity is 51-85% of predicted. For every patient randomly assigned to the placebo group, two will receive pirfenidone. Patients are largely drawn from the Puerto Rican population and are simultaneously enrolled in clinical protocol 95-HG-193. They are admitted to the NIH Clinical Center for 2-3 day admissions every 4 months. The primary efficacy variable is change in forced vital capacity, determined on every admission. Secondary efficacy variables are also examined. A CT scan of the chest and bone densitometry are performed. After 4 years of patient accrual, 35 patients were enrolled; the original statistical analysis plan (SAP) called for 39 patients to be enrolled within one year. The NHGRI DSMB revised the original SAP to perform an interim data analysis 12 months after 30 patients were enrolled, i.e., in May of 2009. That analysis directed the study to stop due to futility. However, this protocol will continue to provide pirfenidone to the three original protocol patients still enrolled, and to any pirfenidone-treated patients who choose to undergo pulmonary lavage to help us determine the effects of pirfenidone on the cytokine profile of alveolar macrophages. The lavages would require enrollment in a separate protocol. The treatment drug will be stopped immediately for all placebo patients and for pirfenidone patients who do not plan to enroll in the lavage protocol. Pirfenidone treatment will stop just after the lavage is performed on patients who do enroll in the lavage protocol, 04-HG-0211. All patients will be invited to continue to come to the NIH annually under the HPS natural history protocol, 95-HG-0193.

ELIGIBILITY:
* INCLUSION CRITERIA

For the portion of the protocol involving continuations of pirfenidone treatment, the criteria are simply previous enrollment in 97-HG-0085.

For enrollment in the new clinical trial, the inclusion criteria involve enrollment in protocol 95-HG-0193, "Clinical and Basic Investigations into Hermansky-Pudlak Syndrome". This itself requires a diagnosis of HPS based upon molecular grounds or the electron microscopic demonstration of deficiency of platelet dense bodies. In addition, for protocol 97-HG-0085, patients must:

* Be over 18 years of age.
* Have an FVC greater than 50 percent and less than or equal to 85 percent of predicted OR a hemoglobin-corrected DL(co) greater than 35 percent and less than or equal to 80 percent of predicted, with no evidence of a pulmonary embolism.
* Have evidence of reduced exercise tolerance lasting longer than one week on either the St. George's Hospital Respiratory Questionnaire or the Dyspnea Perception Scale.
* FEV(1)/FVC greater than 80 percent of predicted after bronchodilators.
* No evidence of improvement in pulmonary fibrosis within the past year defined as an FVC increased by 10 percent or a DL(co) increased by 15 percent.
* Distance walked greater than or equal to 150 meters (492 feet) with oxygen saturation greater than or equal to 83 percent on less than or equal to 6 L/min. of oxygen during the 6-Minute Walk Test (6MWT).
* Be available, willing, and able to come to the NIH Clinical Center for admission every 4 months for three years.

EXCLUSION CRITERIA

* History of clinically significant environmental exposure known to cause pulmonary fibrosis (including but not limited to drugs, asbestos, beryllium, radiation, domestic birds).
* An explanation for interstitial lung disease other than HPS, including but not limited to radiation, sarcoidosis, hypersensitivity pneumonitis, bronchiolitis obliterans organizing pneumonia, cancer.
* Diagnosis of any connective tissue disease including but not limited to scleroderma, systemic lupus erythematosus, rheumatoid arthritis.
* Listing on a lung transplantation waiting list.
* Pregnancy or lactation
* Cigarette smoking in the past 6 months
* History of ethanol abuse or recreational drug use in the past two years
* History of human immunodeficiency virus (HIV) or chronic viral hepatitis infection
* Chronic use of high-dose steroids (greater than 10 mg prednisone/day)
* Prior use of pirfenidone
* Use of any of the following within 28 days of enrollment: investigational therapy, cytotoxic/immunosuppressive agents other than corticosteroids (including but not limited to azathioprine, cyclosphosphamide, methotrexate, cyclosporine); cytokine modulators (including but not limited to etanercept and infliximab); therapies targeted to treat pulmonary fibrosis (including but not limited to D-penicillamine, colchicine, interferon gamma-1b, bosentan, N-acetylcysteine
* Any severe medical complication including but not be limited to uncontrolled seizures, repeated transient ischemic attacks, abnormal mental status, severe ataxia, uncontrolled migraine headaches, diplopia, repeated episodes of syncope, untreated clinical depression, recent myocardial infarction (past 6 months), unstable angina, clinically relevant arrhythmias, uncontrolled hypotension or hypertension (systolic blood pressure less than 80 or greater than 180 mm Hg), myocarditis, hepatomegaly (liver greater than 3 cm below the right costal margin), renal glomerular impairment (creatinine clearance less than 35 ml/min/1.73 m2, pancreatitis, toxic thyroiditis, malignancy (except basal cell carcinoma)
* Medications with a high frequency of life threatening side effects
* Significant laboratory abnormalities, including but not limited to serum potassium less than 3.0 or greater than 5.4 mEq/L, SGPT greater than 100 U/L, CK greater than 700 U/L, hemoglobin less than 9.0 g/dL, platelets less than 70 k/mm3, leucocyte count less than 2.0 k/microliter, or cholesterol greater than 400 mg/dL.
* For women of child bearing age, failure to have an effective method of birth control.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2005-09; Primary Completion 2009-09 (Actual); Study Completion 2016-05-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Anikster Y, Huizing M, White J, Shevchenko YO, Fitzpatrick DL, Touchman JW, Compton JG, Bale SJ, Swank RT, Gahl WA, Toro JR. Mutation of a new gene causes a unique form of Hermansky-Pudlak syndrome in a genetic isolate of central Puerto Rico. Nat Genet. 2001 Aug;28(4):376-80. doi: 10.1038/ng576. PMID 11455388
- [Background] Gahl WA, Brantly M, Kaiser-Kupfer MI, Iwata F, Hazelwood S, Shotelersuk V, Duffy LF, Kuehl EM, Troendle J, Bernardini I. Genetic defects and clinical characteristics of patients with a form of oculocutaneous albinism (Hermansky-Pudlak syndrome). N Engl J Med. 1998 Apr 30;338(18):1258-64. doi: 10.1056/NEJM199804303381803. PMID 9562579
- [Background] Gahl WA, Brantly M, Troendle J, Avila NA, Padua A, Montalvo C, Cardona H, Calis KA, Gochuico B. Effect of pirfenidone on the pulmonary fibrosis of Hermansky-Pudlak syndrome. Mol Genet Metab. 2002 Jul;76(3):234-42. doi: 10.1016/s1096-7192(02)00044-6. PMID 12126938
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_1997-HG-0085.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were enrolled at the NIH Clinical Center between September 2005 to March 2009.
Period: Overall Study
Arm/Group | Pirfenidone | Placebo
Started | 23 | 12
Completed | 6 | 2
Not Completed | 17 | 10
Not completed — Death | 1 | 0
Not completed — Withdrawal by Subject | 3 | 1
Not completed — Study Termination | 12 | 9
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pirfenidone | Placebo | Total
Number analyzed (Participants) | 23 | 12 | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 22 | 12 | 34
  >=65 years | 1 | 0 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.53 (11.00) | 43.97 (8.02) | 41.05 (10.18)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 6 | 21
  Male | 8 | 6 | 14
Region of Enrollment [Number; unit: participants]
  United States | 23 | 12 | 35
Forced Vital Capacity [Mean (Standard Deviation); unit: % of predicted] — Forced Vital Capacity (FVC) is the volume of air that can be forcibly blown out from the lungs after full inspiration. It is recorded as the percentage of predicted volume (predicted FVC volume is calculated based on subject's height, age, sex, and weight). FVC normal range is 80-120% of predicted.
  % of predicted | 72.77 (8.12) | 73.53 (10.09) | 73.03 (8.70)
Total Lung Capacity [Mean (Standard Deviation); unit: % of predicted volume] — Total Lung Capacity (TLC) is the volume in the lungs at maximal inflation. TLC is recorded as the percentage of predicted volume based on subject's height, age, sex, and weight. TLC normal range is 80-120% of predicted.
  % of predicted volume | 73.84 (12.07) | 73.28 (10.09) | 73.65 (11.28)
Adjusted Diffusing Capacity of the Lung for Carbon Monoxide [Mean (Standard Deviation); unit: % of predicted volume] — Adjusted Diffusing Capacity of the lung for carbon monoxide (DLCOa) measures gas uptake during a single inspiration in a standard time, adjusted for subject's hemoglobin levels. DLCOa is recorded as a percentage of predicted volume, and normal range is 75-125% of predicted.
  % of predicted volume | 67.82 (15.94) | 66.83 (16.60) | 67.48 (15.93)
6 Minute Walk Test [Mean (Standard Deviation); unit: meters] — 6 minute walk test (6MWT) measures the distance that a patient can quickly walk on a flat hard surface in a period of six minutes.
  meters | 517.39 (112.79) | 526.87 (103.00) | 520.65 (107.94)

OUTCOME MEASURES:

1. Primary Outcome: Change in Forced Vital Capacity (36 Months)
Description: Change from baseline in the Forced Vital Capacity (FVC) measurement at 36 months. FVC is the volume of air that can be forcibly blown out from the lungs after full inspiration. FVC is recorded as the percentage of predicted volume (predicted FVC volume is calculated based on subject's height, age, sex, and weight).
Time Frame: Measured at baseline and 36 months
Population: Participants from the Intent to Treat population for whom data was available at baseline and 36 months.
Measure: Mean (Standard Deviation); unit: % of predicted volume
Arm/Group | Pirfenidone | Placebo
Number analyzed (Participants) | 11 | 3
% of predicted volume | -23.52 (24.32) | -20.93 (25.59)

2. Secondary Outcome: Change in Forced Vital Capacity (12 Months)
Description: Change from baseline in the Forced Vital Capacity (FVC) measurement at 12 months. FVC is the volume of air that can be forcibly blown out from the lungs after full inspiration. FVC is recorded as the percentage of predicted volume (predicted FVC volume is calculated based on subject's height, age, sex, and weight).
Time Frame: Measured at baseline and 12 months
Population: Participants from the Intent to Treat population for whom data was available at baseline and 12 months.
Measure: Mean (Standard Deviation); unit: % of predicted volume
Arm/Group | Pirfenidone | Placebo
Number analyzed (Participants) | 18 | 12
% of predicted volume | -7.27 (20.48) | -3.55 (21.33)

3. Secondary Outcome: Change in Total Lung Capacity (36 Months)
Description: Change from baseline in Total Lung Capacity (TLC) measured at 36 months. TLC is the volume in the lungs at maximal inflation. TLC is recorded as the percentage of predicted volume based on subject's height, age, sex, and weight.
Time Frame: Measured at baseline and 36 months
Population: Participants from the Intent to Treat population for whom data is available at baseline and 36 months.
Measure: Mean (Standard Deviation); unit: % of predicted volume
Arm/Group | Pirfenidone | Placebo
Number analyzed (Participants) | 11 | 3
% of predicted volume | -25.26 (24.42) | -22.9 (23.69)

4. Secondary Outcome: Change in Total Lung Capacity (12 Months)
Description: Change from baseline in Total Lung Capacity (TLC) measured at 12 months. TLC is the volume in the lungs at maximal inflation. TLC is recorded as the percentage of predicted volume based on subject's height, age, sex, and weight.
Time Frame: Measured at baseline and 12 months
Population: Participants from the Intent to Treat population for whom data was available at baseline and 12 months.
Measure: Mean (Standard Deviation); unit: % of predicted volume
Arm/Group | Pirfenidone | Placebo
Number analyzed (Participants) | 18 | 12
% of predicted volume | -8.96 (21.03) | 0.53 (21.27)

5. Secondary Outcome: Change in Adjusted Diffusing Capacity of the Lung for Carbon Monoxide (36 Months)
Description: Change from baseline in adjusted Diffusing Capacity of the lung for carbon monoxide (DLCOa) measured at 36 months. DLCOa measures gas uptake during a single inspiration in a standard time, adjusted for subject's hemoglobin levels.
Time Frame: Measured at baseline and 36 months
Population: Participants from the Intent to Treat population for whom data was available at baseline and 36 months.
Measure: Mean (Standard Deviation); unit: % of predicted volume
Arm/Group | Pirfenidone | Placebo
Number analyzed (Participants) | 11 | 3
% of predicted volume | -15.25 (29.89) | -14.93 (29.74)

6. Secondary Outcome: Change in Adjusted Diffusing Capacity of the Lung for Carbon Monoxide (12 Months)
Description: Change from baseline in adjusted Diffusing Capacity of the lung for carbon monoxide (DLCOa) measured at 12 months. DLCOa measures gas uptake during a single inspiration in a standard time, adjusted for subject's hemoglobin levels.
Time Frame: Measured at baseline and 12 months
Population: Participants from the Intent to Treat population for whom data is available at baseline and 12 months.
Measure: Mean (Standard Deviation); unit: % of predicted volume
Arm/Group | Pirfenidone | Placebo
Number analyzed (Participants) | 18 | 12
% of predicted volume | -3.11 (26.47) | -4.74 (25.97)

7. Secondary Outcome: Change in 6 Minute Walk Test (36 Months)
Description: Change from baseline of the 6 minute walk test (6MWT) at 36 months. The 6MWT measures the distance that a patient can quickly walk on a flat hard surface in a period of six minutes.
Time Frame: Measured at baseline and 36 months
Population: Participants from the Intent to Treat population for whom data is available at baseline and 36 months.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Pirfenidone | Placebo
Number analyzed (Participants) | 10 | 2
meters | -232.86 (284.26) | -306.75 (314.69)

8. Secondary Outcome: Change in 6 Minute Walk Test (12 Months)
Description: Change from baseline of the 6 minute walk test (6MWT) at 12 months. The 6MWT measures the distance that a patient can quickly walk on a flat hard surface in a period of six minutes.
Time Frame: Measured at baseline and 12 months
Population: Participants from the Intent to Treat population for whom data is available at baseline and 12 months.
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Pirfenidone | Placebo
Number analyzed (Participants) | 16 | 12
meters | -40.56 (192.66) | -17.21 (201.21)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected over the entire period of the double-blind portion of the study, 4 years.
Arm/Group | Pirfenidone | Placebo
Serious Adverse Events (participants affected / at risk) | 6/23 | 2/12
Other Adverse Events (participants affected / at risk) | 18/23 | 9/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pirfenidone (N=23) | Placebo (N=12)
Blood creatinine phosphokinase increased (Investigations) | 1 (1) | 1 (1)
Chest pain (Cardiac disorders) | 2 (2) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 1 (1) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pirfenidone (N=23) | Placebo (N=12)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 2 (2)
Arthalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Chest pain (Cardiac disorders) | 3 (3) | 1 (1)
Dizziness (Nervous system disorders) | 4 (4) | 0 (0)
Drug eruption (Immune system disorders) | 2 (2) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 12 (12) | 6 (6)
Fatigue (General disorders) | 2 (2) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4) | 1 (1)
Palpitations (Cardiac disorders) | 3 (3) | 0 (0)
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 2 (2) | 2 (2)
Somnolence (Nervous system disorders) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 1 (1) | 0 (0)
Urticaria (Immune system disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 2 (2)

LIMITATIONS AND CAVEATS:
Study enrollment progressed more slowly than anticipated (spanning >3 years instead of one). The Data Safety and Monitoring Board performed an interim analysis one year after 30 subjects enrolled and directed the study to stop due to futility.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No